CLINICAL TRIAL: NCT04396015
Title: Evaluating Cognitive and Functional Impairment in Alzheimer's Dementia With a Ketogenic Diet.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Principal Investigator, Angela Juby, Professor of Medicine, University of Alberta
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00054165
Record Dates: First submitted 2017-10-05; First posted 2020-05-20 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Cognitive Function 1, Social

STUDY DESIGN:
Intervention Model Description: randomized, placebo control cross-over study, with an open label extension
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind placebo controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- medium chain triglyceride (MCT) vs placebo (Placebo Comparator): MCT or placebo (olive oil) for 4 months. Crossover at 4 months
  Interventions: Dietary Supplement: Bulletproof Brain Octane; Dietary Supplement: Placebo
- open label extension (Other): 6 months of MCT oil.
  Interventions: Dietary Supplement: Bulletproof Brain Octane

INTERVENTIONS:
Dietary Supplement: Bulletproof Brain Octane — Medium chain triglyceride oil (MCT)
Dietary Supplement: Placebo — Placebo (olive) oil
  Arms: medium chain triglyceride (MCT) vs placebo

SUMMARY:
The present study is being done in a scientifically rigorous manner, using readily available MCT oil (refined from coconut oil) versus a placebo oil to assess any cognitive and functional benefits for AD patients.

DETAILED DESCRIPTION:
The proposed study, is a randomized placebo controlled cross-over study for 6 months, with an open label extension for another 6 months designed to test the benefits and safety of MCT oil in patients with established AD. It will be the first study on MCT oil ever done with this design, and for this duration in AD.

ELIGIBILITY:
Inclusion Criteria:

* Patients >49years with a clinical diagnosis of AD
* Mini Mental Status Examination (MMSE) score 10-29/30
* on stable dose of medications for 3 months (AChEI, memantine and antidepressants allowed)
* able to speak English
* patient or designate able to sign informed consent
* stable chronic medical conditions (Heart disease, thyroid disease)
* reliable caregiver

Exclusion Criteria:

* age <50 years
* medically unstable
* unable to swallow liquids
* diagnosis of diabetes mellitus
* residence in a nursing/long term care home
* allergy to coconut
* allergy to olive oil

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
cognition | 15months
  Mini Mental Status Examination (MMSE). 0-30. Higher score with higher cognitive function
Cognition | 15 months
  Montreal Cognitive Assessment (MoCA) 0-30. Higher score with higher cognition
cognition | 15 months
  Cognigram (Cogstate) 0-200. Higher score with higher cognitive function
Behavior | 15 months
  Neuropsychiatric Inventory (NPI) 0-96 Higher score with more behaviour problems
Function | 15 months
  Katz Activities of Daily Living Scale 0-6 Higher score with poorer ADL function

SECONDARY OUTCOMES:
maximum tolerated daily dose (ml) of MCT oil | 11 months
  tolerability of MCT oil
maximum tolerated daily dose (ml) of placebo (olive) oil | 4 months
  tolerability of placebo oil
Serum cholesterol mmol/l | 15 months
  safety (% change from baseline)
Serum Triglyceride mmol/l | 15 months
  safety (% change from baseline)
Serum Low density lipoprotein (LDL) mmol/l | 15 months
  safety (% change from baseline)
Dual Energy Absorptiometry (DXA) Body fat | 15 months
  safety (% change from baseline)
Incidence of treatment-emergent Adverse events | 15 months
  safety. Mild, moderate or severe events.

IPD SHARING:
Plan to Share IPD: No